CLINICAL TRIAL: NCT00166153
Title: The Relationships Between Mycophenolic Acid Levels, T-Cell Subsets and Outcomes in Pediatric Heat Transplant Recipients Receiving Mycophenolate Mofetil (Cellcept)
Brief Title: Outcomes in Pediatric Heart Transplant Recipients Receiving Cellcept
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kirk R. Kanter, MD, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0685-2002
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Cardiac Transplantation
Keywords: cardiac transplantation; pediatrics; cardiology; drug metabolism
MeSH Terms: interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: Mycophenolate Mofetil

SUMMARY:
The survival of children who have received heart transplants has greatly improved over the last ten years. One reason for this is better control over rejection. Rejection medications require a delicate balance of enough medicine to work without causing side effects. It is a goal to avoid both rejection and side effects from the anti-rejection medicines. Usually several medicines are used together to prevent rejection. One of these medicines is often Mycophenolic Acid or CellceptThis medicine has been used longer for adults than is has for children. More information is needed on using it for children. The dose is usually determined by the patient's weight or body surface area.

There have been some early studies of the use of Cellcept, but none have proven a relationship between the blood level of the drug and how well it works. More also needs to be known about how this drug works with other anti-rejection drugs and how it works in boys and girls. This study will look more closely at proper dosing, how Cellcept works with other anti-rejection medications, side effects, and any differences in how this medicine works in boys and girls.

All patients in the study will be receiving Cellcept and have blood levels of the drug drawn. Results of their usual treatment and testing will be recorded and evaluated for signs of rejection. All the information will be analyzed. Results of this study will be reported to transplant committees locally and nationally.

DETAILED DESCRIPTION:
Pediatric heart transplant recipients receiving MMF will undergo study testing to measure MPA levels by the HPLC method and T-cell subsets by flow cytometry method. As standard of care they receive histological grading of routine endomyocardial biopsies using the International Society of Heart Lung Transplantation (ISHLT) grading scale. The data obtained from standard assessments will include medications, echocardiographic reports, pre-and post biopsy assessments/physical exams, hospital records for any inpatient hospitalization, and any laboratory assessments. Also, information will be collected on all patients which will be examined for tolerance and success (side effects and rejection) of immunosuppressive therapy.

In newly transplanted patients, study testing will occur at the same time as standard of care biopsies which are typically 1 week, 2 weeks, 3 weeks, 4 weeks, 6 weeks, 8 weeks, 3 months, 4 months, 5 months, 6 months, 8 months, 10 months, 12 months. If the patient has additional visits due to rejection or changes in immunosuppression, then more frequent study testing may be done per investigator preference. Previously transplanted patients will have study testing at the same time as their standard of care visits, usually annually.

ELIGIBILITY:
Inclusion Criteria:

* Heart Transplant Recipients who are transplanted during the course of this study.
* Age 2 weeks to 18 years
* Receiving or plan to receive Mycophenolate mofetil therapy
* Patient/Family has signed an informed assent/consent

Exclusion Criteria:

* Patients that are unable to follow protocol schedule of assessment
* Patients with chronic autoimmune disease
* Patients who have received a multiple organ transplant (i.e. heart-liver, heart-lung etc.)

Ages: 2 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2003-01; Study Completion 2005-05

PRIMARY OUTCOMES:
Examine t-cell subsets to determine the correlation between MIP levels and clinical outcome as well as effect on T-cell proliferation.

SECONDARY OUTCOMES:
Examine histologic grading of routine endomyocardial biopsies to determine the correlation between MPS levels and acute rejections.

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Kanter, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] Keck BM, Bennett LE, Rosendale J, Daily OP, Novick RJ, Hosenpud JD. Worldwide thoracic organ transplantation: a report from the UNOS/ISHLT International Registry for Thoracic Organ Transplantation. Clin Transpl. 1999:35-49. PMID 11038624
- [Background] Laks H, Marelli D, Odim J, Fazio D. Heart transplantation in the young and elderly. Heart Fail Rev. 2001 Sep;6(3):221-6. doi: 10.1023/a:1011406022657. PMID 11391040
- [Background] Sarris GE, Smith JA, Bernstein D, Griffin ML, Pitlick PT, Baum D, Billingham ME, Oyer PE, Stinson EB, Starnes VA, et al. Pediatric cardiac transplantation. The Stanford experience. Circulation. 1994 Nov;90(5 Pt 2):II51-5. PMID 7955282
- [Background] Dipchand AI, Pietra B, McCrindle BW, Rosebrook-Bicknell HL, Boucek MM. Mycophenolic acid levels in pediatric heart transplant recipients receiving mycophenolate mofetil. J Heart Lung Transplant. 2001 Oct;20(10):1035-43. doi: 10.1016/s1053-2498(01)00305-9. PMID 11595558
- [Background] Morissette P, Albert C, Busque S, St-Louis G, Vinet B. In vivo higher glucuronidation of mycophenolic acid in male than in female recipients of a cadaveric kidney allograft and under immunosuppressive therapy with mycophenolate mofetil. Ther Drug Monit. 2001 Oct;23(5):520-5. doi: 10.1097/00007691-200110000-00004. PMID 11591897